CLINICAL TRIAL: NCT03008343
Title: Combination of Irreversible Electroporation and NK Immunotherapy for Recurrent Liver Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRE-NK-Liver
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2018-12

CONDITIONS: Recurrent Liver Carcinoma
Keywords: Irreversible Electroporation; NK Immunotherapy; Recurrent Liver Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Electroporation

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Electroporation and natural killer (Experimental): In this group, the patients will receive regular irreversible electroporation (IRE) treatment in combination with multiple natural killer (NK) immunotherapies. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: Irreversible Electroporation; Biological: Natural killer
- Electroporation (Active Comparator): In this group, the patients will receive regular irreversible electroporation (IRE) treatment to control the tumor growth. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Device: Irreversible Electroporation

INTERVENTIONS:
Device: Irreversible Electroporation — One kind of electric ablation machine from Angiodynamic company (USA)
  Other Names: IRE, NanoKnife
Biological: Natural killer — Each treatment: 8-10 billion cells in all, transfuion in 3 times, i.v.
  Other Names: HANK cell
  Arms: Electroporation and natural killer

SUMMARY:
The aim of this study is the safety and efficacy of irreversible electroporation (IRE) plus natural killer (NK) immunotherapy to recurrent liver cancer.

DETAILED DESCRIPTION:
By enrolling patients with recurrent liver cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using IRE and NK cells.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 5 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Relief degree of tumors | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
Overall survival（OS） | 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Fuda cancer institute of Fuda cancer hospital, Guangzhou, Guangdong, China